CLINICAL TRIAL: NCT03175393
Title: Relation Between Postprandial Lipogram and Coronary Artery Disease Severity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, amgad youssef abdo deep, DOCTOR, Assiut University
Other Study IDs: assiutU01
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Postprandial Dyslipidemia
MeSH Terms: interventions — Coronary Angiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- postprandial dyslipidemia
  Interventions: Device: coronary angiography

INTERVENTIONS:
Device: coronary angiography — per cutaneous coronary intervention to identify severity of coronary artery disease by syntx score

SUMMARY:
Coronary artery disease (CAD) is usually used to refer to the pathological problem affecting the coronary arteries (usually atherosclerosis) that leads to Coronary Heart disease (CHD) which includes the diagnoses of angina pectoris, MI and silent myocardial ischemia.

Despite the mortality for this condition has gradually declined over the last decades in western countries, it still causes about one-third of all deaths in people older than 35 years.

Dyslipidemia is very important risk factors of atherosclerosis that is one of the causes leading to cardiovascular disease Despite management of dyslipidemia by controling fasting total plasma cholesterol and LDL cholesterol as these are the best biomarkers for prediction of cardiovascular diseases (CVD) risk.

LDL elevation is absent in many patients with atherosclerosis and about 1/3 of cardiac events remains to be unpredicted using this method. Even more, in fasting normolipidemic subjects, increased CVD risk is associated with an exaggerated postprandial lipemic response.

Postprandial dyslipidemia is defined as a rise in triglyceride-rich lipoproteins (TRLs), including chylomicron remnants (CMRs) and remnant lipoproteins (RLPs), after eating, has drawn an increasing interest recently because of its association with cardiovascular events. Chylomicron remnants (CMRs) have been shown to penetrate the artery wall and to be retained within the intima.

Endothelial dysfunction is an initial process of atherogenesis and it contributes to the pathogenesis of CHD. Postprandial hyperlipidemia (postprandial hypertriglyceridemia) is involved in the production of proinflammatory cytokines, recruitment of neutrophils, and generation of oxidative stress, resulting in endothelial dysfunction

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is usually used to refer to the pathological problem affecting the coronary arteries (usually atherosclerosis) that leads to Coronary Heart disease (CHD) which includes the diagnoses of angina pectoris, MI and silent myocardial ischemia.

Despite the mortality for this condition has gradually declined over the last decades in western countries, it still causes about one-third of all deaths in people older than 35 years.

Dyslipidemia is very important risk factors of atherosclerosis that is one of the causes leading to cardiovascular disease.

Despite management of dyslipidemia by controling fasting total plasma cholesterol and LDL cholesterol as these are the best biomarkers for prediction of cardiovascular diseases (CVD) risk (5).LDL elevation is absent in many patients with atherosclerosis and about 1/3 of cardiac events remains to be unpredicted using this method. Even more, in fasting normolipidemic subjects, increased CVD risk is associated with an exaggerated postprandial lipemic response.

Atherosclerosis is initiated by vascular endothelium dysfunction followed by formation of macrophage foam cells, which is generated by scavenging of lipids from plasma lipoproteins. Accumulation of foam cells and then proliferation of vascular smooth muscle cells (VSMCs) causes the appearance of fatty streaks, the first visible lesions in the vessel wall.

Postprandial dyslipidemia is defined as a rise in triglyceride-rich lipoproteins (TRLs), including chylomicron remnants (CMRs) and remnant lipoproteins (RLPs), after eating, has drawn an increasing interest recently because of its association with cardiovascular events. Chylomicron remnants (CMRs) have been shown to penetrate the artery wall and to be retained within the intima

remnant-like lipoproteins (RLPs) have been found in human atherosclerotic plaque as well.(9,10) CMRs and TRLs have also been demonstrated to cause endothelial dysfunction, macrophage foam cell formation and the proliferation of VSMCs.

Endothelial dysfunction is an initial process of atherogenesis and it contributes to the pathogenesis of CHD. Postprandial hyperlipidemia (postprandial hypertriglyceridemia) is involved in the production of proinflammatory cytokines, recruitment of neutrophils, and generation of oxidative stress, resulting in endothelial dysfunction in healthy subjects, hypertriglyceridemic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented coronary artery disease and stable for 3 months with no secondary dyslipidemia as hypothyroidism and renal impairment

Exclusion Criteria:

* patients with acute coronary syndrome or any cause of Secondary dyslipidemia

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: documented stable coronary artery disease patients submitted to coronary angiography at assiut university catheterization lab
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Relationship of postprandial lipid profile .HDL and coronary artery disease severity | 1 year
  candidates will be subjected to ;
  Full History taking including:
  * history of DM and its management
  * history of hypertension and its management
  * history of drug abuse
  * family history
  Patient Examination as:
  * BMI
  * waist circumference
    -investigations as:
  * ECG
  * Echocardiography
  * lipid profile
  We will check fasting (14 hours fasting) and 2 hours postprandial lipogram after fat loading with 17 g/body surface (m2),then we will assess CAD severity by coronary angiography using syntax score

CONTACTS AND LOCATIONS:
Overall Officials: Hosam Elaraby, MD, Study Chair — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cervellin G, Lippi G. Of MIs and men--a historical perspective on the diagnostics of acute myocardial infarction. Semin Thromb Hemost. 2014 Jul;40(5):535-43. doi: 10.1055/s-0034-1383544. Epub 2014 Jun 26. PMID 24967888
- [Background] Rosamond W, Flegal K, Furie K, Go A, Greenlund K, Haase N, Hailpern SM, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell C, Roger V, Sorlie P, Steinberger J, Thom T, Wilson M, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2008 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2008 Jan 29;117(4):e25-146. doi: 10.1161/CIRCULATIONAHA.107.187998. Epub 2007 Dec 17. No abstract available. PMID 18086926
- [Background] Nichols M, Townsend N, Scarborough P, Rayner M. Cardiovascular disease in Europe 2014: epidemiological update. Eur Heart J. 2014 Nov 7;35(42):2929. doi: 10.1093/eurheartj/ehu378. No abstract available. PMID 25381246
- [Background] Graham I, Atar D, Borch-Johnsen K, Boysen G, Burell G, Cifkova R, Dallongeville J, De Backer G, Ebrahim S, Gjelsvik B, Herrmann-Lingen C, Hoes A, Humphries S, Knapton M, Perk J, Priori SG, Pyorala K, Reiner Z, Ruilope L, Sans-Menendez S, Op Reimer WS, Weissberg P, Wood D, Yarnell J, Zamorano JL, Walma E, Fitzgerald T, Cooney MT, Dudina A, Vahanian A, Camm J, De Caterina R, Dean V, Dickstein K, Funck-Brentano C, Filippatos G, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Altiner A, Bonora E, Durrington PN, Fagard R, Giampaoli S, Hemingway H, Hakansson J, Kjeldsen SE, Larsen ML, Mancia G, Manolis AJ, Orth-Gomer K, Pedersen T, Rayner M, Ryden L, Sammut M, Schneiderman N, Stalenhoef AF, Tokgozoglu L, Wiklund O, Zampelas A; European Society of Cardiology (ESC); European Association for Cardiovascular Prevention and Rehabilitation (EACPR); Council on Cardiovascular Nursing; European Association for Study of Diabetes (EASD); International Diabetes Federation Europe (IDF-Europe); European Stroke Initiative (EUSI); International Society of Behavioural Medicine (ISBM); European Society of Hypertension (ESH); European Society of General Practice/Family Medicine (ESGP/FM/WONCA); European Heart Network (EHN). European guidelines on cardiovascular disease prevention in clinical practice: executive summary. Fourth Joint Task Force of the European Society of Cardiology and other societies on cardiovascular disease prevention in clinical practice (constituted by representatives of nine societies and by invited experts). Eur J Cardiovasc Prev Rehabil. 2007 Sep;14 Suppl 2:E1-40. doi: 10.1097/01.hjr.0000277984.31558.c4. No abstract available. PMID 17726406
- [Background] Proctor SD, Vine DF, Mamo JC. Arterial retention of apolipoprotein B(48)- and B(100)-containing lipoproteins in atherogenesis. Curr Opin Lipidol. 2002 Oct;13(5):461-70. doi: 10.1097/00041433-200210000-00001. PMID 12352009
- [Background] Zilversmit DB. Atherogenesis: a postprandial phenomenon. Circulation. 1979 Sep;60(3):473-85. doi: 10.1161/01.cir.60.3.473. PMID 222498
- [Background] Kadar A, Glasz T. Development of atherosclerosis and plaque biology. Cardiovasc Surg. 2001 Apr;9(2):109-21. doi: 10.1016/s0967-2109(00)00097-1. PMID 11250172
- [Background] Pal S, Semorine K, Watts GF, Mamo J. Identification of lipoproteins of intestinal origin in human atherosclerotic plaque. Clin Chem Lab Med. 2003 Jun;41(6):792-5. doi: 10.1515/CCLM.2003.120. PMID 12880143
- [Background] Rapp JH, Lespine A, Hamilton RL, Colyvas N, Chaumeton AH, Tweedie-Hardman J, Kotite L, Kunitake ST, Havel RJ, Kane JP. Triglyceride-rich lipoproteins isolated by selected-affinity anti-apolipoprotein B immunosorption from human atherosclerotic plaque. Arterioscler Thromb. 1994 Nov;14(11):1767-74. doi: 10.1161/01.atv.14.11.1767. PMID 7947602
- [Background] van Oostrom AJ, Sijmonsma TP, Verseyden C, Jansen EH, de Koning EJ, Rabelink TJ, Castro Cabezas M. Postprandial recruitment of neutrophils may contribute to endothelial dysfunction. J Lipid Res. 2003 Mar;44(3):576-83. doi: 10.1194/jlr.M200419-JLR200. Epub 2002 Dec 16. PMID 12562833
- [Background] Ceriello A, Assaloni R, Da Ros R, Maier A, Piconi L, Quagliaro L, Esposito K, Giugliano D. Effect of atorvastatin and irbesartan, alone and in combination, on postprandial endothelial dysfunction, oxidative stress, and inflammation in type 2 diabetic patients. Circulation. 2005 May 17;111(19):2518-24. doi: 10.1161/01.CIR.0000165070.46111.9F. Epub 2005 May 2. PMID 15867169
- [Background] Tanaka A, Tomie N, Nakano T, Nakajima K, Yui K, Tamura M, Numano F. Measurement of postprandial remnant-like particles (RLPs) following a fat-loading test. Clin Chim Acta. 1998 Jul 6;275(1):43-52. doi: 10.1016/s0009-8981(98)00073-4. PMID 9706842
- [Derived] Razik NA, Deep AY, Abokrisha MZ, Mosad E, Hasan-Ali H. The relationship between lipid profile after fat loading and coronary artery disease severity assessed by SYNTAX score. ARYA Atheroscler. 2022 May;18(5):2416. doi: 10.48305/arya.2022.16286.2416. Epub 2022 Dec 15. PMID 40231017